CLINICAL TRIAL: NCT04296890
Title: SORAYA: A Phase 3, Single Arm Study of Mirvetuximab Soravtansine in Platinum-Resistant, Advanced High-Grade Epithelial Ovarian, Primary Peritoneal, or Fallopian Tube Cancers With High Folate Receptor-Alpha Expression
Brief Title: A Study of Mirvetuximab Soravtansine in Platinum-Resistant, Advanced High-Grade Epithelial Ovarian, Primary Peritoneal, or Fallopian Tube Cancers With High Folate Receptor-Alpha Expression
Acronym: SORAYA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: ImmunoGen, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IMGN853-0417; 2020-000179-19 (EudraCT Number)
Record Dates: First submitted 2020-02-27; First posted 2020-03-05 (Actual); Results first posted 2024-08-07 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-07

CONDITIONS: Epithelial Ovarian Cancer; Peritoneal Cancer; Fallopian Tube Cancer
Keywords: Platinum resistant; Folate-receptor alpha expression; Phase 3; Antibody-drug conjugate; mirvetuximab soravtansine; IMGN853; Epithelial Ovarian Cancer; Peritoneal Cancer; Fallopian Tube Cancer; MIRV; FRα
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial; Fallopian Tube Neoplasms | interventions — mirvetuximab soravtansine

STUDY DESIGN:
Intervention Model Description: All participants will receive single-agent MIRV at 6 mg/kg adjusted ideal body weight (AIBW) administered on Day 1 of every 3-week cycle (Q3W)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): All participants will receive single-agent mirvetuximab soravtansine (MIRV) at 6 mg/kg adjusted ideal body weight (AIBW) administered on Day 1 of every 3-week cycle (Q3W).
  Interventions: Drug: Mirvetuximab Soravtansine

INTERVENTIONS:
Drug: Mirvetuximab Soravtansine — Mirvetuximab Soravtansine is an antibody drug conjugate designed to target folate receptor α (FRα). It consists of the humanized anti-FRα mAb M9346A attached via a cleavable disulfide linker to the cytotoxic maytansinoid, DM4.
  Other Names: IMGN853; MIRV

SUMMARY:
This study is designed to evaluate the efficacy and safety of mirvetuximab soravtansine (MIRV) in participants with platinum-resistant high-grade serous epithelial ovarian cancer, primary peritoneal, or fallopian tube cancer, whose tumors express a high-level of Folate Receptor-Alpha (FRα). Participants will be, in the opinion of the Investigator, appropriate for single-agent therapy for their next line of therapy. All participants will receive single-agent MIRV at 6 mg/kg adjusted ideal body weight administered on Day 1 of every 3-week cycle.

DETAILED DESCRIPTION:
This study is designed to evaluate the efficacy and safety of mirvetuximab soravtansine (MIRV) in participants with platinum-resistant high-grade serous epithelial ovarian cancer, primary peritoneal, or fallopian tube cancer, whose tumors express a high-level of Folate Receptor Alpha (FRα). Participants will be, in the opinion of the Investigator, appropriate for single-agent therapy for their next line of therapy. FRα positivity will be defined by the Ventana FOLR1 (Folate Receptor 1/Folate Receptor Alpha) Assay.

Approximately 110 eligible participants will be enrolled to achieve a total of 105 efficacy evaluable participants. Efficacy evaluable participants include those who have measurable lesions per Response Evaluation Criteria in Solid Tumors, version 1.1 (RECIST v1.1) at baseline and received at least 1 dose of MIRV.

All participants will receive single-agent MIRV at 6 mg/kg adjusted ideal body weight (AIBW) administered on Day 1 of every 3-week cycle (Q3W).

Tumor response will be evaluated by the Investigator using RECIST v1.1. Computerized tomography (CT) or magnetic resonance imaging (MRI) scans will be collected for sensitivity analysis by blinded independent central review (BICR).

Participants will continue to receive MIRV until disease progression, unacceptable toxicity, withdrawal of consent, death, or until the Sponsor terminates the study (whichever comes first).

Tumor assessments, including radiological assessments by CT/MRI scans will be performed at Screening and subsequently every 6 weeks (± 1 week) from Cycle 1 Day 1 (C1D1) for the first 36 weeks then every 12 weeks (± 3 weeks) until disease progression, death, the start of new anticancer therapy, or participant's withdrawal of consent (whichever occurs first).

Participants who discontinue MIRV for reasons other than progressive disease (PD) will continue with tumor assessments until documentation of PD or the start of a new anticancer therapy, whichever comes first. Prior to Week 36 (from Cycle 1, Day 1), assessments should occur every 6 weeks (± 1 week) as allowed by local requirements but must occur at an interval of no more than 12 weeks. After Week 36, assessment will occur every 12 weeks (± 3 weeks) until documentation of PD or the start of new anticancer therapy.

All participants who discontinue MIRV will be followed for survival every 3 months (± 1 month) until death, lost to follow-up, withdrawal of consent for survival follow-up, or end of study (EOS) (whichever comes first). Additional survival follow-up calls may occur periodically, if needed.

ELIGIBILITY:
Inclusion Criteria:

1. Female participants ≥ 18 years of age
2. Participants must have a confirmed diagnosis of high-grade serous epithelial ovarian cancer (EOC), primary peritoneal cancer, or fallopian tube cancer
3. Participants must have platinum-resistant disease:

   1. Participants who have only had 1 line of platinum based therapy must have received at least 4 cycles of platinum, must have had a response (complete response/remission [CR] or partial response/remission [PR]) and then progressed between > 3 months and ≤ 6 months after the date of the last dose of platinum
   2. Participants who have received 2 or 3 lines of platinum therapy must have progressed on or within 6 months after the date of the last dose of platinum

   Note: Progression should be calculated from the date of the last administered dose of platinum therapy to the date of the radiographic imaging showing progression

   Note: Participants who are platinum refractory during front-line treatment are excluded (see exclusion criteria)
4. Participants must have progressed radiographically on or after their most recent line of anticancer therapy.
5. Participants must be willing to provide an archival tumor tissue block or slides, or undergo procedure to obtain a new biopsy using a low-risk, medically routine procedure for immunohistochemistry (IHC) confirmation of Folate Receptor α (FRα) positivity
6. Participant's tumor must be positive for FRα expression as defined by the Ventana FOLR1 Assay
7. Participants must have at least 1 lesion that meets the definition of measurable disease by RECIST v1.1 (radiologically measured by the Investigator)
8. Participants must have received at least 1 but no more than 3 prior systemic lines of anticancer therapy, including at least 1 line of therapy containing bevacizumab, and for whom single-agent therapy is appropriate as the next line of treatment:

   1. Adjuvant ± neoadjuvant considered 1 line of therapy
   2. Maintenance therapy (e.g., bevacizumab, poly adenosine diphosphate-ribose polymerase (PARP) inhibitors) will be considered part of the preceding line of therapy (i.e., not counted independently)
   3. Therapy changed due to toxicity in the absence of progression will be considered part of the same line (i.e., not counted independently)
   4. Hormonal therapy will be counted as a separate line of therapy unless it was given as maintenance
9. Participants must have an Eastern Cooperative Oncology Group Performance Status (ECOG PS) of 0 or 1
10. Participants must have completed prior therapy within the specified times below:

    1. Systemic antineoplastic therapy within 5 half-lives or 4 weeks (whichever is shorter) prior to first dose of MIRV
    2. Focal radiation completed at least 2 weeks prior to first dose of MIRV
11. Participants must have stabilized or recovered (Grade 1 or baseline) from all prior therapy-related toxicities (except alopecia)
12. Participants must have completed any major surgery at least 4 weeks prior to first dose of MIRV and have recovered or stabilized from the side effects of prior surgery
13. Participants must have adequate hematologic, liver and kidney functions defined as:

    1. Absolute neutrophil count (ANC) ≥ 1.5 x 10^9/L (1,500/μL) without G-CSF in the prior 10 days or long-acting WBC growth factors in the prior 20 days
    2. Platelet count ≥ 100 x 10^9/L (100,000/μL) without platelet transfusion in the prior 10 days
    3. Hemoglobin ≥ 9.0 g/dL without packed red blood cell (PRBC) transfusion in the prior 21 days
    4. Serum creatinine ≤ 1.5 x upper limit of normal (ULN)
    5. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 3.0 x ULN
    6. Serum bilirubin ≤ 1.5 x ULN (patients with documented diagnosis of Gilbert syndrome are eligible if total bilirubin < 3.0 x ULN)
    7. Serum albumin ≥ 2 g/dL
14. Participants or their legally authorized representative must be willing and able to sign the informed consent form (ICF) and to adhere to the protocol requirements
15. Women of childbearing potential (WCBP) must agree to use highly effective contraceptive method(s) while on MIRV and for at least 3 months after the last dose
16. WCBP must have a negative pregnancy test within the 4 days prior to the first dose of MIRV

Exclusion Criteria:

1. Male participants
2. Participants with endometrioid, clear cell, mucinous, or sarcomatous histology, mixed tumors containing any of the above histologies, or low-grade/borderline ovarian tumor
3. Participants with primary platinum-refractory disease, defined as disease that did not respond to (CR or PR) or has progressed within 3 months of the last dose of first-line platinum-containing chemotherapy
4. Participants with prior wide-field radiotherapy (RT) affecting at least 20 percent of the bone marrow
5. Participants with > Grade 1 peripheral neuropathy per Common Terminology Criteria for Adverse Events (CTCAE)
6. Participants with active or chronic corneal disorders, history of corneal transplantation, or active ocular conditions requiring ongoing treatment/monitoring, such as uncontrolled glaucoma, wet age-related macular degeneration requiring intravitreal injections, active diabetic retinopathy with macular edema, macular degeneration, presence of papilledema, and /or monocular vision
7. Participants with serious concurrent illness or clinically relevant active infection, including, but not limited to the following:

   1. Active hepatitis B or C infection (whether or not on active antiviral therapy)
   2. Human immunodeficiency virus (HIV) infection
   3. Active cytomegalovirus infection
   4. Any other concurrent infectious disease requiring IV antibiotics within 2 weeks prior to the first dose of MIRV

   Note: Testing at screening is not required for the above infections unless clinically indicated
8. Participants with a history of multiple sclerosis (MS) or other demyelinating disease and/or Lambert-Eaton syndrome (paraneoplastic syndrome)
9. Participants with clinically significant cardiac disease including, but not limited to, any of the following:

   1. Myocardial infarction ≤ 6 months prior to first dose
   2. Unstable angina pectoris
   3. Uncontrolled congestive heart failure (New York Heart Association > class II)
   4. Uncontrolled ≥ Grade 3 hypertension (per CTCAE)
   5. Uncontrolled cardiac arrhythmias
10. Participants with a history of hemorrhagic or ischemic stroke within 6 months prior to enrollment
11. Participants with a history of cirrhotic liver disease (Child-Pugh Class B or C)
12. Participants with a previous clinical diagnosis of noninfectious interstitial lung disease (ILD), including noninfectious pneumonitis
13. Participants requiring use of folate-containing supplements (eg, folate deficiency)
14. Participants with prior hypersensitivity to monoclonal antibodies (mAb)
15. Women who are pregnant or breastfeeding
16. Participants who received prior treatment with MIRV or other FRα-targeting agents
17. Participants with untreated or symptomatic central nervous system (CNS) metastases
18. Participants with a history of other malignancy within 3 years prior to enrollment.

    Note: Participants with tumors with a negligible risk for metastasis or death (eg, adequately controlled basal-cell carcinoma or squamous-cell carcinoma of the skin, or carcinoma in situ of the cervix or breast) are eligible
19. Prior known hypersensitivity reactions to study drugs and/or any of their excipients

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 106 (Actual)
Dates: Start 2020-07-23 (Actual); Primary Completion 2021-11-16 (Actual); Study Completion 2022-11-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Method, MD, MPH, MBA, Study Director — ImmunoGen, Inc.; Ursula Matulonis, MD, Principal Investigator — Dana-Farber Cancer Institute; Robert Coleman, MD, Principal Investigator — The US Oncology Network
Locations (89):
- United States (34):
  - Arizona Oncology Associates, Phoenix, Arizona
  - City of Hope Medical Center, Duarte, California
  - California Cancer Associates (cCARE), Fresno, California
  - Stanford School of Medicine, Palo Alto, California
  - California Pacific Medical Center Research Institute, San Francisco, California
  - Rocky Mountain Cancer Centers, Littleton, Colorado
  - Sarasota Memorial Health Care System, Sarasota, Florida
  - Florida Cancer Specialists Panhandle, Tallahassee, Florida
  - University of South Florida, Tampa, Florida
  - Florida Cancer Specialists Research, West Palm Beach, Florida
  - Northside Hospital, Atlanta, Georgia
  - Hinsdale Hospital, Hinsdale, Illinois
  - St. Vincent Gynecologic Oncology, Indianapolis, Indiana
  - University of Kansas Cancer Center, Westwood, Kansas
  - Norton Cancer Institute, Louisville, Kentucky
  - Women's Cancer Center, Covington, Louisiana
  - Maryland Oncology Hematology, P.A., Rockville, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Midwest Oncology Associates/Sarah Cannon, Kansas City, Missouri
  - Center of Hope at Renown Medical Center, Reno, Nevada
  - Holy Name Medical Center, Teaneck, New Jersey
  - Mount Sinai Health System, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Sarah Cannon Research Institute / Tennessee Oncology, PLLC, Nashville, Tennessee
  - Texas Oncology-Austin Central, Austin, Texas
  - Texas Oncology, P.A. - Fort Worth Cancer Center, Fort Worth, Texas
  - Texas Oncology, P.A. - McAllen, McAllen, Texas
  - Texas Oncology, P.A. - Sugar Land, Sugar Land, Texas
  - USOR: Texas Oncology - The Woodlands, Gynecologic Oncology, The Woodlands, Texas
  - Texas Oncology, P.A. - Tyler, Tyler, Texas
  - Kadlec Clinic Hematology and Oncology, Kennewick, Washington
  - University of Wisconsin Carbone Cancer Center, Madison, Wisconsin
  - Froedtert and the Medical College of Wisconsin Department of Obstetrics & Gynecology, Milwaukee, Wisconsin
- Australia (4):
  - Royal North Shore Hospital, St Leonards, New South Wales
  - ICON Cancer Care, Auchenflower, Queensland
  - Peninsula and South Eastern Haematology & Oncology Group, Frankston, Victoria
  - St John of God Subiaco Hospital, Subiaco, Western Australia
- Belgium (5):
  - Cliniques Universitaires Saint Luc - lnstitut Roi Albert II, Brussels, Brussels Capital
  - Centre Hopsitalier de l'Ardenne, Libramont, Luxembourg
  - UZ Gent, Ghent
  - UZ Leuven, Leuven
  - CHU UCL Namur/Site Sainte Elisabeth, Namur
- MHAT "Serdika", Sofia, Bulgaria
- Všeobecná fakultní nemocnice v Praze, Prague, Prague, Czechia
- Germany (3):
  - Universitätsmedizin Mannheim, Mannheim, Baden-Wurttemberg
  - UMG Frauenklinik Robert-Koch-Str. 40, Göttingen, Lower Saxony
  - KEM, Essen
- Ireland (6):
  - Mater Misericordiae University Hospital, Dublin, Leinster
  - St. James's Hospital, Dublin, Leinster
  - Cork University Hospital, Cork, Munster
  - Bon Secours Hospital, Cork, Munster
  - University Hospital Waterford, Waterford, Munster
  - Beaumont Hospital, Dublin
- Israel (7):
  - Rambam Medical Center, Haifa
  - Shaare Zedek Medical Center, Jerusalem
  - Hadassah Ein Kerem Medical center, Jerusalem
  - Meir Medical Center, Kfar Saba
  - Sheba Medical Center, Ramat Gan
  - Kaplan Medical Center, Rehovot
  - Ziv Medical Center, Safed
- Italy (10):
  - Policlinico S. Orsola-Malpighi, Bologna
  - Azienda Socio Santaria Territoriale degli Spedali Civili di Brescia, Brescia
  - Istituto Oncologico Candiolo, Candiolo
  - Ospedale Cannizzaro di Catania, Catania
  - IEO Istituto Europeo di Oncologia, Milan
  - Azienda Ospedaliera Ospedale Niguarda Ca'Granda, Milan
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Napoli
  - Istituto Nazionale Tumori- G. Pascale, Napoli
  - Ospedale S.Maria della Misericordia, Perugia
  - Fondazione Policlinico Universitario A. Gemelli IRCCS, Roma
- Poland (3):
  - Specjalistyczna Przychodnia Lekarska Medicus, Chorzów, Silesian Voivodeship
  - Mazurskim Centrum Onkologiiw Olsztynie, Olsztyn, Warmian-Masurian Voivodeship
  - Instytut Centrum Zdrowia Matki Polki, Lodz, Łódź Voivodeship
- Spain (15):
  - Institut Català d'Oncologia Badalona Hospital Universitari Germans Trias i Pujol, Badalona, Barcelona
  - Hospital La Paz, Madrid, Castellana
  - Hospital Teresa Herrera - Complejo Hospitalario Universitario A Coruna, A Coruña, Galicia
  - Hospital Quirón Dexeus, Barcelona
  - Vall d'Hebron Institute of Oncology, Barcelona
  - lnstitut Catala d' Oncologia L' Hospitalet, Barcelona
  - Hospital Reina Sofia de Cordoba, Córdoba
  - Institut Català d'Oncología de Girona, Girona
  - Clinica Universidad de Navarra, Madrid
  - MD Anderson Cancer Centre, Madrid
  - Hospital Clínico Universitario San Carlos, Madrid
  - Hospital Clinico Universitario Virgen de la Arrixaca, Murcia
  - Corporació Sanitaria Parc Taulí, Sabadell
  - Hospital Clinico Universitario de Valencia, Valencia
  - Instituto Valenciano de Oncologia, Valencia

REFERENCES:
- [Derived] Coleman RL, Lorusso D, Oaknin A, Cecere SC, Denys H, Colombo N, van Gorp T, Konner JA, Romeo Marin M, Harter P, Murphy C, Wang Y, Esteves B, Method M, Matulonis U. Mirvetuximab soravtansine in folate receptor alpha (FRalpha)-high platinum-resistant ovarian cancer: final overall survival and post hoc sequence of therapy subgroup results from the SORAYA trial. Int J Gynecol Cancer. 2024 Aug 5;34(8):1119-1125. doi: 10.1136/ijgc-2024-005401. PMID 38858103
- [Derived] Dilawari A, Shah M, Ison G, Gittleman H, Fiero MH, Shah A, Hamed SS, Qiu J, Yu J, Manheng W, Ricks TK, Pragani R, Arudchandran A, Patel P, Zaman S, Roy A, Kalavar S, Ghosh S, Pierce WF, Rahman NA, Tang S, Mixter BD, Kluetz PG, Pazdur R, Amiri-Kordestani L. FDA Approval Summary: Mirvetuximab Soravtansine-Gynx for FRalpha-Positive, Platinum-Resistant Ovarian Cancer. Clin Cancer Res. 2023 Oct 2;29(19):3835-3840. doi: 10.1158/1078-0432.CCR-23-0991. PMID 37212825
- [Derived] Matulonis UA, Lorusso D, Oaknin A, Pignata S, Dean A, Denys H, Colombo N, Van Gorp T, Konner JA, Marin MR, Harter P, Murphy CG, Wang J, Noble E, Esteves B, Method M, Coleman RL. Efficacy and Safety of Mirvetuximab Soravtansine in Patients With Platinum-Resistant Ovarian Cancer With High Folate Receptor Alpha Expression: Results From the SORAYA Study. J Clin Oncol. 2023 May 1;41(13):2436-2445. doi: 10.1200/JCO.22.01900. Epub 2023 Jan 30. PMID 36716407

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were enrolled at 39 sites in North America, Europe, and Asia Pacific.
Groups:
- Mirvetuximab Soravtansine: Participants received single-agent mirvetuximab soravtansine (MIRV) at 6 milligrams (mg)/kilogram (kg) adjusted ideal body weight (AIBW) administered intravenously (IV) on Day 1 of every 3-week cycle (Q3W).
Period: Overall Study
Arm/Group | Mirvetuximab Soravtansine
Started | 106
INV Efficacy Evaluable Population | 105
Completed | 38
Not Completed | 68
Not completed — Withdrawal by Subject | 1
Not completed — Death | 62
Not completed — Lost to Follow-up | 3
Not completed — Other than specified | 2

BASELINE CHARACTERISTICS:
Population: The Safety population was defined as participants who received at least 1 dose of study drug.
Groups:
- Mirvetuximab Soravtansine: Participants received single-agent mirvetuximab soravtansine (MIRV) at 6 mg/kg AIBW administered IV on Day 1 of every 3-week cycle (Q3W).
Arm/Group | Mirvetuximab Soravtansine
Number analyzed (Participants) | 106
Age, Continuous [Mean (Standard Deviation); unit: years] | 62 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 106
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 99
  Unknown or Not Reported | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 102
  More than one race | 0
  Unknown or Not Reported | 2

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR): Percentage of Participants With Objective Response as Assessed by the Investigator Using Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1)
Description: ORR was defined as percentage of participants with a confirmed best overall response (BOR) of complete response (CR) or partial response (PR). CR: Disappearance of all target or non-target lesions. All pathological or non-pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 millimeters (mm). PR: At least 30% decrease in the sum of the longest diameters (SoD) of target lesions, taking as reference the baseline SoD.
Time Frame: Up to approximately 15 months
Population: The investigator (INV) Efficacy Evaluable population was defined as all participants who received at least 1 dose of study drug and who had measurable disease at baseline by investigator assessment per RECIST 1.1.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Mirvetuximab Soravtansine
Number analyzed (Participants) | 105
percentage of participants | 32.4 [23.6 to 42.2]

2. Secondary Outcome: Duration of Response (DOR) as Assessed by the Investigator Using RECIST v1.1
Description: DOR was defined as the time from the date of the first response (CR or PR), until the date of progressive disease (PD) or death from any cause, whichever occurred first. DOR for participants who had not progressed or died at the time of analysis was censored at the date of their last tumor assessment. PD: At least a 20% increase in the SoD of target lesion, taken as reference the smallest (nadir) SoD since and including baseline. In addition to the relative increase of 20%, the SoD must also demonstrate an absolute increase of at least 5 mm. Unequivocal progression of non-target lesions. Unequivocal progression should not normally trump target lesion status. It must be representative of overall disease status change, not a single lesion increase. DOR was estimated using the Kaplan-Meier method.
Time Frame: Up to approximately 15 months
Population: All participants that showed a CR or PR according to RECIST 1.1 were analyzed.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Mirvetuximab Soravtansine
Number analyzed (Participants) | 34
months | 6.93 [5.55 to 9.66]

3. Secondary Outcome: Percentage of Participants With CA-125 Confirmed Clinical Response Per Gynecologic Cancer Intergroup (GCIG) Criteria
Description: The GCIG CA-125 response was defined as at least 50% reduction in CA-125 levels from baseline. The response must have been confirmed and maintained for at least 28 days.
Time Frame: Up to approximately 15 months
Population: The CA-125-Evaluable population was defined as all participants who received at least 1 dose of study drug and whose pretreatment sample was ≥2.0 times the upper limit of normal (ULN), within 2 weeks prior to first dose of mirvetuximab soravtansine, and who had at least 1 postbaseline CA-125 evaluation.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Mirvetuximab Soravtansine
Number analyzed (Participants) | 86
percentage of participants | 46.5 [35.7 to 57.6]

4. Secondary Outcome: Progression-Free Survival (PFS) as Assessed by the Investigator Using RECIST v1.1
Description: PFS was defined as the time from initiation of study drug until the date of PD or death whichever occurred first, estimated using the Kaplan-Meier method. PD: At least a 20% increase in the SoD of target lesion, taken as reference the smallest (nadir) SoD since and including baseline. In addition to the relative increase of 20%, the SoD must also demonstrate an absolute increase of at least 5 mm. Unequivocal progression of non-target lesions and appearance of new lesions. Unequivocal progression should not normally trump target lesion status. It must be representative of overall disease status change, not a single lesion increase.
Time Frame: Up to approximately 15 months
Population: INV Efficacy Evaluable population was defined as all participants who received at least 1 dose of study drug and who had measurable disease at baseline by investigator assessment per RECIST 1.1.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Mirvetuximab Soravtansine
Number analyzed (Participants) | 105
months | 4.27 [3.71 to 5.22]

5. Secondary Outcome: Overall Survival Assessed by the Investigator Using RECIST v1.1
Description: Overall survival was defined as the time from the date of first dose until the date of death from any cause, estimated using the Kaplan-Meier method.
Time Frame: Up to approximately 27 months
Population: as for outcome 4
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Mirvetuximab Soravtansine
Number analyzed (Participants) | 105
months | 15.0 [11.5 to 18.7]

6. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: An adverse event (AE) was defined as any untoward medical occurrence that develops or worsens in severity during the conduct of a clinical study and does not necessarily have a causal relationship to study drug. TEAEs were defined as AEs with an onset date on or after the first dose of Study drug, and within 30 days of the last dose of study drug or prior to the start of a new anticancer treatment, whichever occurred first. A summary of all Serious Adverse Events (SAEs) and Other Adverse Events (nonserious) regardless of causality is located in the 'Reported Adverse Events' Section.
Time Frame: Up to approximately 27 months
Population: The Safety population was defined as participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Mirvetuximab Soravtansine
Number analyzed (Participants) | 106
Participants | 105

ADVERSE EVENTS:
Time Frame: Up to approximately 27 months
Description: Deaths (all-cause) were assessed from first dose until death (survival follow-up). Serious and nonserious AEs (Safety population) were assessed from first dose and within 30 days of the last dose or prior to the start of a new anticancer treatment, whichever occurred first.
Arm/Group | Mirvetuximab Soravtansine
All-Cause Mortality (participants affected / at risk) | 62/106
Serious Adverse Events (participants affected / at risk) | 36/106
Other Adverse Events (participants affected / at risk) | 102/106
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Mirvetuximab Soravtansine (N=106)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Vasculitis (Vascular disorders) | 1
Administration site extravasation (General disorders) | 1
Disease progression (General disorders) | 1
General physical health deterioration (General disorders) | 1
Malaise (General disorders) | 1
Pyrexia (General disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Substance-induced psychotic disorder (Psychiatric disorders) | 1
Ankle fracture (Injury, poisoning and procedural complications) | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 1
Atrial fibrillation (Cardiac disorders) | 1
Brain stem syndrome (Nervous system disorders) | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1
Anaemia (Blood and lymphatic system disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Ascites (Gastrointestinal disorders) | 5
Colitis microscopic (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Intestinal haemorrhage (Gastrointestinal disorders) | 1
Intestinal obstruction (Gastrointestinal disorders) | 2
Intestinal perforation (Gastrointestinal disorders) | 1
Large intestinal obstruction (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 1
Oesophagitis (Gastrointestinal disorders) | 1
Small intestinal obstruction (Gastrointestinal disorders) | 5
Cholecystitis (Hepatobiliary disorders) | 1
Cholecystitis acute (Hepatobiliary disorders) | 1
Cholestasis (Hepatobiliary disorders) | 1
Hepatitis (Hepatobiliary disorders) | 1
Clostridium difficile infection (Infections and infestations) | 1
Device related infection (Infections and infestations) | 1
Peritonitis bacterial (Infections and infestations) | 1
Severe protein calorie malnutrition (Metabolism and nutrition disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Mirvetuximab Soravtansine (N=106)
Alanine aminotransferase increased (Investigations) | 12
Aspartate aminotransferase increased (Investigations) | 16
Blood alkaline phosphatase increased (Investigations) | 12
Gamma-glutamyltransferase increased (Investigations) | 13
Weight decreased (Investigations) | 6
Dysgeusia (Nervous system disorders) | 8
Headache (Nervous system disorders) | 10
Neuropathy peripheral (Nervous system disorders) | 19
Anaemia (Blood and lymphatic system disorders) | 14
Neutropenia (Blood and lymphatic system disorders) | 16
Thrombocytopenia (Blood and lymphatic system disorders) | 10
Asthenia (General disorders) | 22
Fatigue (General disorders) | 32
Oedema peripheral (General disorders) | 6
Cataract (Eye disorders) | 21
Dry eye (Eye disorders) | 30
Eye pain (Eye disorders) | 9
Keratopathy (Eye disorders) | 34
Photophobia (Eye disorders) | 17
Punctate keratitis (Eye disorders) | 9
Vision blurred (Eye disorders) | 49
Abdominal distension (Gastrointestinal disorders) | 13
Abdominal pain (Gastrointestinal disorders) | 26
Abdominal pain upper (Gastrointestinal disorders) | 13
Ascites (Gastrointestinal disorders) | 6
Constipation (Gastrointestinal disorders) | 32
Diarrhoea (Gastrointestinal disorders) | 33
Dyspepsia (Gastrointestinal disorders) | 6
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 8
Nausea (Gastrointestinal disorders) | 41
Vomiting (Gastrointestinal disorders) | 20
Cough (Respiratory, thoracic and mediastinal disorders) | 7
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 11
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 9
Erythema (Skin and subcutaneous tissue disorders) | 6
Arthralgia (Musculoskeletal and connective tissue disorders) | 17
Back pain (Musculoskeletal and connective tissue disorders) | 8
Myalgia (Musculoskeletal and connective tissue disorders) | 11
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6
Urinary tract infection (Infections and infestations) | 10
Decreased appetite (Metabolism and nutrition disorders) | 20
Hypokalaemia (Metabolism and nutrition disorders) | 11
Hypomagnesaemia (Metabolism and nutrition disorders) | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2020-08-28): https://cdn.clinicaltrials.gov/large-docs/90/NCT04296890/Prot_000.pdf
  • Statistical Analysis Plan (2021-11-05): https://cdn.clinicaltrials.gov/large-docs/90/NCT04296890/SAP_001.pdf